CLINICAL TRIAL: NCT06101953
Title: The Impact of Coping Strategies on Interoception and Psychological Resilience in Response to Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatma Rana Aydemir, Occupational therapist, Hacettepe University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: HU23INSPIRE; E-68552689-000-00003048522 (Other: Hacettepe University Ethics Comission)
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Stress
Keywords: stress; resilience; interoception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Stress management

INTERVENTIONS:
Behavioral: Stress management — It spanned 12 weeks, with three hours per week (comprising two hours of theoretical content and one hour of practical application) and employed diverse teaching methods, including lectures, interactive learning, research, fieldwork, hands-on practice, and question-answer sessions. The primary objective of this course was to enhance students' awareness of stress by helping them identify its sources, symptoms, and effects. Also interception and resilience. Furthermore, it aimed to teach students how to assess stress and apply stress-management techniques effectively in their daily lives.
  Arms: Intervention

SUMMARY:
The goal of this observational study is to explore the impact of a 12-week online knowledge-sharing program focusing on stress management, psychological resilience, and interoception in university students who face various stressors. The primary questions it aims to answer are:

* How does participating in the online program influence students' understanding and management of stress?
* Can engaging in this program enhance students' resilience in the face of academic and life challenges?
* Does the program improve students' interoception skills, helping them recognize and manage internal bodily sensations and emotions more effectively?

Participants will be asked to:

* Attend weekly sessions covering topics such as stress, its sources, stages, diseases related to stress, coping methods, psychological resilience, and interoception.
* Engage in discussions, self-reflection, and practical exercises.
* Share their experiences and insights.
* Complete assessments to measure their perceived stress level, resilience, and interoceptive awareness.

Researchers will compare the group that participates in the program with a control group to determine if the program significantly improves stress management, enhances psychological resilience, and bolsters interoception skills among university students.

DETAILED DESCRIPTION:
Participants and Sampling: The study sample consisted of university students enrolled in the Department of Occupational Therapy at Hacettepe University Faculty of Health Sciences, particularly those taking the Stress Coping Methods course. The determination of the sample size was guided by a rigorous statistical approach, employing G Power for power analysis. Following this, randomization was performed to create both a control group and an intervention group. The inclusion criteria required participants to be at least 18 years old, studying at a university in Turkey, and having Turkish as their native language. The sole exclusion criterion was the presence of any psychiatric diagnosis, ensuring the homogeneity of the sample.

Study Procedure: The intervention program, stretching over 12 weeks, was based on the Stress Coping Mechanisms lecture, derived from various resources such as Pendleton and Schultz-Khron (2001), Brown et al. (2019), and Reitz et al. (2020). Delivered by a seasoned practitioner with over 20 years of expertise in stress coping education, the program consisted of three hours per week. The curriculum was thoughtfully structured to ensure a comprehensive understanding of stress, its sources, stages, diseases associated with stress, coping strategies, psychological resilience, and interoception.

The online knowledge-sharing format encouraged interactivity, with participants engaging in discussions, self-reflection, and practical exercises. As part of the learning process, students were encouraged to conduct self-inquiries and present their findings to the class. The program aimed to provide students with a profound understanding of stress, emphasizing the critical role of psychological resilience and interoception in effective stress management and overall well-being.

Statistical Analysis: The statistical analysis was carried out using SPSS v26 software. The Kolmogorov-Smirnov test was used to assess the normality of all variables. Descriptive statistics were applied, including frequency, percentage, mean, minimum, maximum, and standard deviation for categorical and numerical variables. To evaluate differences between categorical variables, the chi-square test was employed. The Wilcoxon signed-rank test was used to compare baseline and final scores, while the Mann-Whitney U test compared the results between the control and intervention groups. The significance level was set at p<0.05. Detailed statistical analyses were guided by a predefined analytical plan that encompassed both primary and secondary objectives as outlined in the study protocol. Quality assurance, data validation, and other registry-specific procedures were followed in line with best practices, ensuring data integrity and the accuracy of the results. Site monitoring and auditing, data checks for data quality, and source data verification were integral parts of the quality assurance plan. Additionally, a data dictionary containing detailed variable descriptions, as well as Standard Operating Procedures for various registry operations, was meticulously maintained. Further components included sample size assessment, a plan for addressing missing data, and a comprehensive statistical analysis plan to address the primary and secondary objectives as specified in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over 18 years of age.
* Participants must speak and understand the Turkish language fluently.
* Participants must be enrolled in the Stress Coping Methods course at Hacettepe University.

Exclusion Criteria:

* Participants with any psychiatric diagnosis were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-06-11 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Level | 12 weeks
  The Perceived Stress Scale (PSS), a self-report questionnaire, is used to measure participants' perceived stress in various life situations. It consists of 14 items that assess the extent to which specific situations in an individual's life are perceived as stressful. Participants evaluate each item on a 5-point Likert scale, ranging from "Never (0)" to "Very Often (4)."

SECONDARY OUTCOMES:
Interoceptive Sensory Questionnaire | 12 weeks
  Interoceptive awareness was assessed using the Interoceptive Sensory Questionnaire, which is a self-report questionnaire designed to evaluate individuals' ability to perceive internal sensory information. The questionnaire consists of items inquiring about how individuals feel and interpret sensory cues from their bodies, with responses scored on a scale from 1 to 7. The scale defines individuals scoring 71 and above as "Alexithymia," and those scoring 94 and above as "High Alexithymia."
Brief Resilience Scale | 12 weeks
  Psychological resilience was assessed using the Brief Resilience Scale (BRS). The BRS is a 5-item self-report scale designed to measure individuals' psychological resilience. The scale uses a 5-point Likert format, and after reverse-coding certain items, higher scores on the BRS indicate greater psychological resilience. Adaptation of the scale to Turkish, as well as the validation and reliability study, were conducted by Doğan (2015).

CONTACTS AND LOCATIONS:
Overall Officials: Onur Altuntas, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy and confidentiality concerns.